CLINICAL TRIAL: NCT07159529
Title: Flapless Versus Flap Technique for Evaluation of Crestal Bone Loss and Osseointegration of Dental Implants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Abdalla Mohammed Faqe Wais, principal investigator, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OS 3-24-2165
Record Dates: First submitted 2025-08-29; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Posterior Mandible Missing Tooth and /or Teeth
Keywords: flap and flapless dental implant insertion techniques

STUDY DESIGN:
Intervention Model Description: participants of this study trial were divided into two groups,a group of them received dental implants with flapless technique and the other group of participants received dental implants with conventional flap elevation technique.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- flapless group (Experimental): 10 patients received dental implants just by taking a punch of tissue
  Interventions: Procedure: flapless technique; Procedure: tissue punching
- flap group (Experimental): conventional flap elevation to place dental imp;lant
  Interventions: Procedure: flap technique

INTERVENTIONS:
Procedure: flapless technique — taking a punch of tissue to place dental implant through surgical guide
  Arms: flapless group
Procedure: flap technique — conventional flap elevation and drilling to place dental implant
  Arms: flap group
Procedure: tissue punching — just a punch of tissue taken to place dental implant
  Arms: flapless group

SUMMARY:
this study aimed to evaluate both clinically and radiographically the effect of flapless versus flap techniques on initial crestal bone loss and osseointegration of dental implants in lower posterior area. the study is to designed to observe the clinical outcomes such as primary stability and pain within initial hours and days and secondary stability over a 6 month period .

DETAILED DESCRIPTION:
this clinical trial was designed to observe the clinical outcomes of techniques of implant installation including flapless and flap techniques about their effect on; osseointegration that measured by checking dental implants stability with resonance frequency analysis device after 6 months of their installation, initial crestal bone loss around the dental implants after 6 months of their installation that that evaluated radiographically and also recording pain perception by the patients within the initial hours and days after implant insertion by both techniques.The patients collected and operated from department of Oral and Maxillofacial surgery, Faculty of Dentistry, Tanta University, Egypt.

Approval of this research was obtained from Faculty of Dentistry, Tanta University Research Ethics Committee (REC). The purpose of the present study was explained to the patients and informed consents were obtained according to the guidelines on human research published by the REC at Faculty of Dentistry, Tanta University.

ELIGIBILITY:
Inclusion Criteria:

Patients that fulfill one or more of the following criteria were included:

1. Residual bone height of alveolar ridge more than 8 mm.
2. Residual bone width of alveolar ridge more than 4 mm.
3. Healthy and sufficient covering soft tissue (keratinized mucosa).
4. Distance between inferior border of mandible and the crest of alveolar ridge more than 2cm.
5. Motivated, cooperative patients with good oral hygiene.

Exclusion criteria:

1. Patients with relevant systemic disorder that may compromise bone healing (e.g.: Uncontrolled diabetic).
2. Extraction socket less than 4 months of healing time.
3. Patient with Autoimmune disease, or neurologic disorder.
4. Heavy smokers (more than 15 cigarettes/day).93
5. Bad oral hygiene.
6. Patients with history of radiotherapy or chemotherapy.
7. Patients who are fully edentulous.

Exclusion Criteria:

-

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-05-23 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
crestal bone loss and osseointegration | 6 months postoperatively
  initial crestal bone loss around the dental implants measured radiographically and secondary stability checked after six months to check osseointegration of the dental implants by resonance frequency analysis device.

CONTACTS AND LOCATIONS:
Overall Officials: Marwa Taha Ibrahim, Assistant Professor, Principal Investigator — faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Gharbia Governorate, Egypt